CLINICAL TRIAL: NCT06150248
Title: Effect of Health Education Intervention on Promoting Healthy Lifestyles for Undergraduate Female Students at Northern Border University in Saudi Arabia
Brief Title: Effect of Health Education Intervention on Promoting Healthy Lifestyles for Undergraduate Female Students in Saudi Arabia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Putra Malaysia (Other)
Collaborators: Northern Border University (Other)
Responsible Party: Principal Investigator, Hanan Alzarea, Principal Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: UPM-PhD Hanan
Record Dates: First submitted 2023-11-20; First posted 2023-11-29 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Obesity; Physical Inactivity
MeSH Terms: conditions — Obesity; Sedentary Behavior | interventions — Early Intervention, Educational

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial (RCT) design
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Other): Intervention group: Participants assigned to the intervention group will receive educational intervention program to improve their knowledge and promote lifestyle adherence in terms of healthy diet behaviour and physical activity among the undergraduate students. This program will include educational booklets and educational classes include six weeks of in-person education sessions and six weeks of social media messaging. The course will include six weekly teaching units (lectures and group discussions, 45-60 minutes each):
  Topic 1: To understand the causes and prevention strategies for overweight and obesity.
  Topic 2: To understand food based approaches to reduce or prevent overweight and obesity.
  Topic 3: To understand the importance of regular physical activity. Topic 4: To demonstrate how snacking can be a healthy habit. Topic 5: To learn how to read and interpret food labels. Topic 6: To understand how to prepare healthy meals.
  Interventions: Other: Education Intervention
- Control group: No Intervention (Other): Participants randomized to the control group in this study will not receive any intervention (They will have their regular curriculums and normal physical activity routine).
  Interventions: Other: No intervention

INTERVENTIONS:
Other: Education Intervention — This intervention is based on the Social Cognitive Theory (SCT) and The Health Belief Model (HBM) to improve knowledge and promote lifestyle adherence in terms of healthy diet behaviour and physical activity among the undergraduate students. This program will include educational booklets and educational classes include six weeks of in-person education sessions and six weeks of social media messaging. The course will include six weekly teaching units (lectures and group discussions, 45-60 minutes each):
  Topic 1: To understand the causes and prevention strategies for overweight and obesity.
  Topic 2: To understand food based approaches to reduce or prevent overweight and obesity.
  Topic 3: To understand the importance of regular physical activity. Topic 4: To demonstrate how snacking can be a healthy habit. Topic 5: To learn how to read and interpret food labels. Topic 6: To understand how to prepare healthy meals.
  Arms: Intervention group
Other: No intervention — They will have their regular curriculums and normal physical activity routine.
  Arms: Control group: No Intervention

SUMMARY:
According to the World Health Organization (WHO), Saudi Arabia has seen a more astonishing rise in obesity. Young females have a considerable prevalence of unhealthy dietary practices and lack of knowledge about healthy and energy-dense foods. Additionally, in Saudi Arabia, the levels of physical inactivity ranged from about one-third to as high as 70% of the population. The current study aims to determine the effects of combined health education and motivational message intervention on promoting healthy lifestyles and body composition markers for undergraduate female students who suffer from obesity at Northern Border University in the Kingdom of Saudi Arabia.

DETAILED DESCRIPTION:
A cluster randomized controlled study will be conducted among 250 undergraduate female students aged (18-24) in Northern Border University. The intervention and control faculties will be selected and allocated randomly. The intervention group will have six weeks of fortnightly six sessions (45 minutes), while the control group will have their regular curriculums and normal physical activity routine. The research instruments include socio-demographic characteristics, anthropometric measurements, and questionnaires about knowledge, attitude, and practice of obesity, physical activity, dietary intake, dietary quality, diet and eating behaviour, and disordered eating. Data will be collected from intervention and control groups at baseline, post-intervention, and 3-month follow-up after the intervention. Data will be analyzed by using the (SPSS) software version 26. Descriptive statistics will be used to distribute and summarize the data. A Generalized Estimating Equation (GEE) will be used to test the effect of the intervention program for the selected variables (outcomes) between and within the group at baseline, six weeks, and one month after intervention, which is adjusted for clustering.

ELIGIBILITY:
Inclusion Criteria:

* Female undergraduate students.
* Saudi students.
* Aged between 18-24 years.
* Categorized with a BMI greater than 25.

Exclusion Criteria:

* Pregnant students
* Students with diseases on treatment such as asthma, diabetes, cancer, cardiovascular diseases, fractures, cirrhosis, or other diseases.
* Students with any medical condition who not allowed to do physical activity.

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only Female undergraduate students.
Enrollment: 250 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
1. Improve Knowledge, Attitude and Practice of Obesity | [Time Frame: Timepoint 1 = Baseline. Repeated measurement: Timepoint 2 = week 12 (12-week post-intervention)]]
  The knowledge, attitude, and practice of obesity will be measured using a self-report instrument knowledge, attitudes, and practices questionnaire (KAPQ) modified by Laar et al. (2020). The questionnaire will consist of close-ended questions divided into three sections: The knowledge section will cover participants' understanding of obesity, its causes, consequences, and prevention strategies. The attitudes section will capture participants' feelings and opinions towards overweight obesity. Some of the items under this section will include how participants feel about their body shape, weight, and diet. The last section will capture participants' practices related to obesity, including the frequency of consumption of fast foods, sweets, refined carbohydrate foods, vegetables, and fruits.
2. Change the Body mass index (BMI) | [Time Frame: Timepoint 1 = Baseline. Repeated measurement: Timepoint 2 = week 12 (12-week post-intervention)]]
  The Body mass index (BMI) will be report in kg/m^2 by using the following formula (BMI = kg/m2 where kg is a person's weight in kilograms and m2 is their height in metres squared). Body weight will be measured using Omron HBF 375 to the nearest 0.1 kg. SECA body meter 206 will be employed to measure their heights to the nearest 0.1 cm. Body mass index (BMI) will be classified into (underweight, normal weight, overweight, and obesity). If the BMI is less than 18.5, it falls within the underweight range. If the BMI is 18.5 to <25, it falls within the healthy weight range. If the BMI is 25.0 to <30, it falls within the overweight range. If the BMI is 30.0 or higher, it falls within the obesity range.

SECONDARY OUTCOMES:
3. Improve the Physical Activity. | [Time Frame: Timepoint 1 = Baseline. Repeated measurement: Timepoint 2 = week 12 (12-week post-intervention)]]
  The Physical Activity will be measured using a self-report instrument international physical activity questionnaire (IPAQ). The IPAQ was determined to be reliable (Craig et al., 2003) and valid (Lee et al., 2011). It uses the types of intensity of physical activity and sitting time that people do as part of their daily lives to estimate the total physical activity per week and time spent sitting. The IPAQ has seven open-ended questions surrounding the individuals' last 7-day recall of vigorous, moderate and sedentary physical activities; frequency (in days per week) and duration (time per day). Participants in the both groups will respond to the IPAQ at three points of the study (beginning, post-intervention and 3-month follow-up).
4. Change Dietary Intake, Dietary Quality, Diet and Eating Behavioural | [Time Frame: Timepoint 1 = Baseline. Repeated measurement: Timepoint 2 = week 12 (12-week post-intervention)]]
  The dietary intake, dietary quality and eating behaviour will be measured by using a self-report instrument a Saudi food frequency questionnaire (SFFQ). The SFFQ captures the frequency of consumption (number of times per week) and quantity of foods consumed (serving sizes) by participants over the past 12 months. It includes 140 food items that include a variety of meats, bread and cereals, sandwiches and burgers, dairy products, sweets and meats, drinks, fruits and vegetables. The questionnaire has 61 questions related to food consumption. In addition, a 24-hour dietary recall (24HR-DR) questionnaire will be used. The participants will name all foods consumed in the past 24 hours, the source of foods, the quantities of foods, method of preparation as well as the time of the day the foods were consumed.
5. Improve Disordered Eating | [Time Frame: Timepoint 1 = Baseline. Repeated measurement: Timepoint 2 = week 12 (12-week post-intervention)]]
  The disordered eating will be measured by using a self-report instrument Eating attitude test 26 (EAT-26) a questionnaire. The questionnaire comprised 2 main sections including the Eating attitude test 26 to measured weight concerns and abnormal eating. Also, including an additional 5 eating behaviors questions.
6. Change Sedentary Activity | [Time Frame: Timepoint 1 = Baseline. Repeated measurement: Timepoint 2 = week 12 (12-week post-intervention)]]
  Sedentary Activity will be measured by using a self-report instrument the Sedentary Activity Questionnaire (SAQ). The questionnaire will ask the participants how many hours and minutes they spent in eleven different sedentary behaviours per day on weekdays and weekends. The questionnaire classified the eleven sedentary behaviours into five categories (Screen time, education, travel, cultural activities and social activities). Participants indicate high sedentary behaviour if the total time of (SAQ) 4 hrs/day, while < 4 hrs/day means low sedentary behaviour.

CONTACTS AND LOCATIONS:
Overall Officials: Geeta Appannah, PhD, Study Chair — Department of Nutrition , Faculty of Medicine and Health Sciences, UniversitI Putra Malaysia (UPM), 43400 Serdang, Selangor, Malaysia
Locations (1):
- Geeta Appannah, Serdang, Selangor, Malaysia